CLINICAL TRIAL: NCT04939675
Title: Modification of Epilepsy Screen Questionnaire and Treatment Feasibility Evaluation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202104076MINA
Record Dates: First submitted 2021-06-15; First posted 2021-06-25 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Zonisamide; Levetiracetam; Lamotrigine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anti-seizure medication (Experimental): The intervention group will receive anti-epileptic drug treatment according to the guideline of American Epilepsy Society 15 for 12 weeks. The recommended regimens include zonisamide, lamotrigine, or levetiracetam at the minimal therapeutic doses (zonisamide 100mg twice daily, levetiracetam 500mg twice daily, lamotrigine 50mg twice daily), and the choices depend on tolerability of the participants and contraindications (allergy to any drugs, or allergy to sulphonamides in zonisamide users). The participants will be followed every 4 weeks.
  Interventions: Drug: Zonisamide 100mg; Drug: Levetiracetam 500mg; Drug: LamoTRIgine 50mg
- Observation (No Intervention): The participants will be followed every 4 weeks without anti-seizure medication.

INTERVENTIONS:
Drug: Zonisamide 100mg — Only one ASM will be used. The drug choice depends on patients tolerance and basic condition. Twice daily
  Other Names: Zonegran 100mg
  Arms: Anti-seizure medication
Drug: Levetiracetam 500mg — Only one ASM will be used. The drug choice depends on patients tolerance and basic condition. Twice daily
  Other Names: Keppra 500mg
  Arms: Anti-seizure medication
Drug: LamoTRIgine 50mg — Only one ASM will be used. The drug choice depends on patients tolerance and basic condition. Twice daily
  Other Names: Lamictal 50mg
  Arms: Anti-seizure medication

SUMMARY:
Atypical presentations in epilepsy may include confusion status, acute maniac or delirious condition, loss of cognitive ability such as speech, interaction skills, or other praxis. Current diagnosis of epilepsy did not address on definition of seizure. The new insights of seizure semiology and their treatment response, suggest the screen tool and diagnostic criteria of epilepsy can be revised.

In this study, we have two aims. The first aim is to develop a screening questionnaire by adding new semiology of epilepsy, including abnormality in psychiatry, cognition, and sleep, and to test its accuracy. The second aim is to evaluate the benefits in cognition of anti-epileptic drug intervention in participants with positive screening results.

DETAILED DESCRIPTION:
The age-adjusted prevalence and incidence of epilepsy were 5.85 (per 1,000) and 97 (per 100,000 person-years) in Taiwan according to a database survey from National Health Insurance. In community screen of 13,663 subjects aged 30 years or older in Keelung, 52 patients were found with epilepsy, which corresponded to a 2.77/1000 of prevalence rate. Of those patients, 24.3% had never been diagnosed before.

The screening of epilepsy was based on questionnaires, including questions inquiring whether the patients have motor manifestation of epilepsy, including motor convulsion, twitching (myoclonus), behavior arrest, sudden falling, loss of consciousness, or known diagnosis of epilepsy. Recently, literature has reported atypical initial presentation of epilepsy such as rapid cognitive decline and mood disturbance. A study of patients with severe psychiatric disorders has also found that 1.6% cases had undiagnosed epilepsy, which was higher than that in general population. Atypical presentations in epilepsy may include confusion status, acute maniac or delirious condition, loss of cognitive ability such as speech, interaction skills, or other praxis. Additionally, vomiting, terrors, or hyperkinetic movements during sleep may also be observed in patients with epilepsy. Indeed, the International League Against Epilepsy has included cognitive, emotional, and sensory as non-motor onset presentations in its new classification.

The diagnosis of epilepsy was based on any at least two unprovoked (or reflex) seizures occurring >24 h apart. However, the diagnosis did not address on definition of seizure. Anti-seizure medications (ASMs) had been reported to improve cognitive performance in the older people with cognitive impairment and epileptiform discharge on electroencephalography. There was also a report of recovery of long-term anterograde amnesia after initiation of an ASM in a case of transient epileptic amnesia. The new insights of seizure semiology and their treatment response, suggest the screen tool and diagnostic criteria of epilepsy can be revised.

In this study, we have two aims. The first aim is to develop a screening questionnaire by adding new semiology of epilepsy, including abnormality in psychiatry, cognition, and sleep, and to test its accuracy. We used the 9-question screening questionnaire as a backbone. Additional questions included Q10: sleep events including sleep-onset vomiting, night scare, or hyperkinetic movement paroxysmal cognitive events (Q11: any paroxysmal agitation or confusion; Q12: any paroxysmal function loss, including communication, praxis, or other mental function); rapid progressive events (Q13: rapid progressive cognitive decline; Q14: recent hallucination, delusion, change in mood and behaviors). The questionnaire will then be translated into traditional Chinese version by a bilingual qualified neurologist. The translated version will then back-translated into English by an independent bilingual researcher and will finally be determined by a group of experts in neuropathy, pain, and linguistics.

The second aim is to evaluate the benefits in cognition of anti-epileptic drug intervention in participants with positive screening results. After excluding participants with diagnosis of epilepsy per criteria as above, participants are recruited to the antiepileptic drug trial if they fulfill positive responses in Q11-Q14 of the questionnaire or the Mini-Mental State Examination (MMSE) ≦ 24, and presence of epileptiform discharge in electroencephalography (EEG), including spikes, sharp waves, temporal intermittent rhythmic delta activity, or other focal or generalized slow waves that could not be explained by physiological or anatomical pathology. Participants who fulfill criteria will be included in this open-labeled randomized study to test efficacy of anti-seizure medication (ASM) in these patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age equal or more than 20-year-old 2a. Patients already diagnosed of epilepsy 2b. Non-epileptic patients from outpatient and inpatient settings of National Taiwan University Hospital (NTUH) and National Taiwan University Hospital Yunlin Branch (NTUHYL) 2c. Community health people

Exclusion Criteria:

1. Participants with cognitive decline (Clinical dementia rating > 1) and could not answer the questionnaire reliably. However, participants will be recruited if their caregivers are fully aware of their recent condition and will help to complete the questionnaire.
2. Pregnancy or breast-feeding
3. Having adverse effect to all the anti-epileptic drug used in the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Mini-Mental State Examination | 12 weeks
  The Mini-Mental State Examination is a common analysis of cognitive function, with a score range from 0 to 30, and higher score indicates a better performance of cognition. We hypothesized that differences after ASM intervention will have a difference score of 4 in comparison to the observational group.

SECONDARY OUTCOMES:
Pattern changes in electroencephalography | 12 weeks
  Changes in electroencephalography, including presence or absence of epileptiform discharges or power of slow(theta and delta) waves will be documented.
Neuropsychiatric Inventory Questionnaire | 12 weeks
  Neuropsychiatric Inventory Questionnaire measures behavior and emotional abnormality, which are rated within a domain in terms of both frequency (1=rarely, less than once per week; 2=sometimes, about once per week; 3=often, several times per week; and 4=very often, once or more per day) and severity (1=mild; 2=moderate; 3=severe), thus yielding a composite symptom domain score (frequency × severity) ranging from 0 (absence of behavioral symptoms) to 144 points (maximum severity of behavioral symptoms).

CONTACTS AND LOCATIONS:
Overall Officials: Kai-Chieh Chang, M.D., Principal Investigator — National Taiwan University Hospital

IPD SHARING:
Plan to Share IPD: No